CLINICAL TRIAL: NCT00346892
Title: Reactogenicity & Immunogenicity Study of Two Doses of GSK Biologicals' Oral Live Attenuated HRV Vaccine Co-administered With Either OPV or IPV in Healthy Infants (Approximately 5-10 Weeks Old) in South Africa
Brief Title: To Evaluate 2 Doses of GSK Biologicals' Oral Live Attenuated Human HRV Vaccine Co-administered With Either OPV or IPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/014
Record Dates: First submitted 2006-02-03; First posted 2006-06-30 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Rotavirus Infections
Keywords: Prophylaxis rotavirus
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines

INTERVENTIONS:
Biological: Rotavirus (vaccine)

SUMMARY:
"The primary objective of this study was to demonstrate that co-administering HRV vaccine with OPV does not induce a significant decrease in poliovirus immune response one month after the third dose of combined vaccines.

The primary objective was reached if one month after the third dose of polio vaccine, upper limit of the 95% CI for the difference in Seroprotection rate between the group B and C pooled and (minus) the group A was below 10% for each polio serotype."

DETAILED DESCRIPTION:
The study had three groups: Group A: HRV + OPV + DTPa/Hib; Group B: HRV + placebo OPV + DTPa-IPV/Hib; Group C: HRV Placebo + OPV + DTPa/Hib. Two cohorts: Subjects enrolled before the 2002 RV season were to receive two doses of HRV or placebo at approximately 6 and 10 weeks of age (first cohort) and subjects enrolled after the 2002 RV season received vaccinations at approximately 10 and 14 weeks of age (second cohort). Routine EPI vaccinations were to be administered concomitantly with the study vaccines.

ELIGIBILITY:
Inclusion criteria: Healthy infants between 5 and 10 weeks of age at first study vaccination with (after the 2002 RV season) confirmed negative HIV status of the subject's mother during pregnancy or thereafter. Exclusion criteria: History of allergic disease, any confirmed or suspected immunosuppressive or immunodeficient condition, clinically significant history of chronic gastrointestinal disease or other serious medical condition as determined by the investigator or had not received treatment prohibited by the protocol.

Ages: 5 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450
Dates: Start 2001-11; Primary Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Seroprotection for each polio serotype 1 month after the 3rd dose.

SECONDARY OUTCOMES:
Proportion of subjects with vaccine take 1 month after each dose of study vaccine, viral shedding in a subset of subjects, presence of RV in diarrheal stools, anti-rota IgA antibody seroconversion rate and serum anti-rota IgA antibody concent

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register